CLINICAL TRIAL: NCT04232657
Title: Romosozumab to Improve Bone Mineral Density and Architecture in Chronic SCI
Acronym: Chronic Romo
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Kessler Institute for Rehabilitation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B3415-R; BAU-19-66 (Other: JJP VAMC Local IRB); 1600530 (Other: JJP VAMC Local IRB); NCT05180032 (obsolete NCT alias)
Record Dates: First submitted 2019-11-25; First posted 2020-01-18 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injury (=3 Years); Sublesional Bone Loss Secondary to SCI
Keywords: Spinal Cord Injury; Veterans Affairs RR&D; Sublesional Bone Loss
MeSH Terms: conditions — Spinal Cord Injuries | interventions — romosozumab; Denosumab; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel group clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and study investigators / team members will be blinded to the treatment group assignment. The designated study drug administrator will be the only individual unblinded. This individual will administer the drug/placebo saline injections behind a sheet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Romosozumab Treatment (baseline to month 11) (Experimental): Of the thirty-nine (39) individuals with chronic spinal cord injury (SCI) enrolled in this study, twenty-six (26) participants will be randomly selected to received romosozumab (210mg SQ) once a month for 12 months.
  Interventions: Drug: Romosozumab
- Placebo (baseline to month 12) (Placebo Comparator): Of the thirty-nine (39) individuals with chronic SCI enrolled in this study, thirteen (13) participants will be randomly selected to received placebo injections (NS SQ) once a month for 12 months. They will follow study procedures identical to those performed by individuals in the treatment (romosozumab) group.
  Interventions: Drug: Placebo
- Denosumab (month 12 to month 24) (Active Comparator): Both groups (treatment and placebo) will receive denosumab (60mg SQ) at months 12 and 18 for maintenance of or to further increase bone mineral density (BMD) at regions of interest (ROI).
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Romosozumab — 39 subjects with chronic SCI will be studied with a 2:1 ratio of randomization of drug to placebo. Romosozumab (210mg SQ) will be administered once a month for 12 months. Participants will arrive at the JJPVAMC or KIR once a month to receive injections of romosozumab or placebo. A designated unblinded healthcare professional will be responsible for administering these injections.
  Other Names: Evenity
  Arms: Romosozumab Treatment (baseline to month 11)
Drug: Denosumab — Because there is a high likelihood that the bone accrued while on romosozumab will be lost once discontinued, denosumab, an anti-resorptive agent, will be administered after treatment with romosozumab, to maintain or, possibly, to continue to increase, bone mineral density. Denosumab will be administered to both groups (treatment and placebo) for an additional 12 months. Participants will be asked to arrive at the JJPVAMC once every 6 months to receive injections of denosumab by a healthcare professional.
  Other Names: Prolia
  Arms: Denosumab (month 12 to month 24)
Drug: Placebo — Thirteen (13) of the thirty-nine (39) subjects enrolled in this study will be randomly selected to receive placebo (NS SQ) injections for 12 months (baseline - month 11). The placebo injections will be administered by an unblinded healthcare professional (registered nurse / physician). Participants will be blinded to their group assignment (romosozumab treatment or placebo).
  Other Names: Normal Saline (NS) injection
  Arms: Placebo (baseline to month 12)

SUMMARY:
Treatment for sublesional bone loss (osteoporosis) in persons with chronic, motor-complete spinal cord injury (SCI) has been limited and unsuccessful to date. Romosozumab, a sclerostin antagonist, has potential to increase bone formation (anabolic) and decrease bone resorption (anti-catabolic) in persons with chronic SCI. Conventional anti-resorptive therapy alone would not be anticipated to reverse sublesional bone loss in a timely manner because the skeleton below the level of lesion in chronic SCI is assumed to be in a low turnover state. However, because there is a high likelihood that the bone accrued while on romosozumab will be lost once discontinued, denosumab, an anti-resorptive agent, will be administered after treatment with romosozumab, to maintain or, possibly, to continue to increase, bone mineral density (BMD).

The purpose of this study is to address the gap in the treatment of osteoporosis in individuals with chronic SCI by partially restoring BMD with romosozumab treatment for 12 months and then to maintain, or further increase, BMD with denosumab treatment for 12 months. A two group, randomized, double-blind, placebo-controlled clinical trial will be conducted in 39 participants who have chronic (>3 years), motor-complete or incomplete SCI and areal BMD (aBMD) values at the distal femur of at the distal femur <1.0 g/cm2 measured by dual photon X-ray absorptiometry (DXA). The intervention group will receive 12 months of romosozumab followed by 12 months of denosumab, and the control group will receive 12 months of placebo followed by 12 months denosumab.

DETAILED DESCRIPTION:
Persons with chronic spinal cord injury (SCI) have markedly reduced bone mass and the loss of skeletal architectural integrity, which predisposes them to low-impact fractures. Currently, there is no practical treatment to reverse the severe bone loss in persons with chronic SCI. In the proposed study, a dual pharmacological intervention will be tested to improve bone health. Restoration of bone mass below the level of injury would be expected to reduce the morbidity associated with fractures and permit safer participation in upright activities. Quality of life would be substantially improved because of the ability to engage more securely in activities of daily living and to integrate into the community. Despite the depressed skeletal activity below the level of lesion in persons with chronic SCI, net bone loss occurs because resorption exceeds formation, with a difference between these rates in those with SCI being greater than that observed in the able-bodied population. Thus, it would be anticipated to be of value in persons with chronic SCI to increase bone turnover with the objective to increase bone formation over that of bone resorption. In a preclinical study that administered an anti-sclerostin antibody to rats 12 weeks after complete spinal cord transection bone, mineral density (BMD) was almost fully restored at the distal femoral metaphysis, with improved bone structure, and mechanical strength; in contrast, vehicle-treated animals after complete spinal transection had a marked reduction in distal femoral metaphysis BMD and a deterioration in bone structure and mechanical strength. When used to treat postmenopausal osteoporosis, romosozumab, a human monoclonal anti-sclerostin antibody, was more effective to increase bone mineral density (BMD) and to reduce fracture than any other anti-resorptive or bone-anabolic agent, and this effect was also evident for the appendicular skeleton, which is the site in individuals with chronic SCI of greatest bone loss and most frequent fracture. Because of the absence of clinical options available for the treatment of osteoporosis in individuals with chronic paralysis, the investigators have proposed to test an antagonist of sclerostin, which is a potent bone anabolic agent with proven efficacy in treating women with postmenopausal osteoporosis, to improve bone mass and reduce fragility fractures.

Thirty-nine male and female subjects with chronic, motor-complete or incomplete SCI (>3 years post injury, American Spinal Injury Association Impairment Scale A & B) between the ages of 18 and 55 years old (for females) or 65 years old (for males) who have aBMD at the distal femur at the distal femur <1.0 g/cm2 will be recruited for participation in a randomized, double-blind, placebo-controlled, parallel group clinical trial. The outcome measures of the proposed study are bone mineral density (BMD) by peripheral quantitative computed tomography (pQCT) and dual energy x-ray absorptiometry (DXA), and biochemical markers of bone resorption and formation. This prospective, randomized, placebo controlled clinical trial will take place at the James J. Peters VA Medical Center (JJPVAMC) and Kessler Institute for Rehabilitation (KIR) (each facility will perform patient enrollment and study procedures).

ELIGIBILITY:
Inclusion Criteria:

* Motor-complete or incomplete SCI [all levels of lesion] classified using International Standards for Neurological Classification for Spinal Cord Injury (ISNCSCI) impairment scale] as ISNCSCI score A-C
* Duration of injury >3 years
* Males (18-65 years old) and females (premenopausal, between the ages of 18 and 55 years old).
* aBMD at the distal femur <1.0 g/cm2 (determined at screening)

Exclusion Criteria:

* Long-bone fracture of the leg within the past year
* History of prior bone disease (Paget's hyperparathyroidism, etc.)
* Active and/or history of coronary heart disease or stroke within the past year
* Postmenopausal women
* Men with known hypogonadism prior to SCI
* Anabolic therapy longer than six months duration after SCI
* Glucocorticoid administration longer than three months duration within the last year, and/or prescribed moderate or high dose corticosteroids (>40 mg/d prednisone or an equivalent dose of other corticosteroid medication) for longer than one week, not including drug administered to preserve neurological function at the time of acute SCI
* Endocrinopathies (hyperthyroidism, Cushing's disease or syndrome, etc.)
* Severe underlying chronic disease (e.g., COPD, end-stage heart disease, chronic renal failure)
* Heterotopic ossification (HO) of the knee region (the distal femoral epiphysis is the primary endpoint); HO to any other boney region will not prevent study participation as long as contraindicated medications have not been prescribed)
* Chronic alcohol abuse
* Hypocalcemia
* Pregnancy
* Prescribed a bisphosphonate for HO, or prescribed any other agent to treat osteoporosis other than calcium and vitamin D
* Electrical stimulation of the lower extremities
* Current diagnosis of cancer or history of cancer
* Osteosarcoma
* Life expectancy less than 5 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-02-05 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in vBMD at the Distal Femur, measured by pQCT after 12 months of romosozumab treatment | Baseline (0), Month 6, Month 12
  Percent change of volumetric BMD (vBMD) (mg/cm^3)at the distal femur, measured by peripheral quantitative computed tomography (pQCT) (slice thickness 2.4mm, default voxel size of 0.5mm), with 12 months of romosozumab therapy. vBMD measurements will be taken at baseline, month 6 and month 12.
Change in vBMD at the distal femur after an additional 12 months of denosumab treatment | Month 18, Month 24
  Percent change of Integral vBMD (mg/cm^3)at the distal femur, measured by pQCT (slice thickness 2.4mm, default voxel size of 0.5mm), after additional 12 months of denosumab therapy. vBMD measurements will be taken by pQCT at months 18 and 24.

OTHER OUTCOMES:
Additional variables by pQCT - vBMD Proximal Tibia | Baseline (0), Month 6, Month 12, Month 18, Month 24
  Percent change in proximal tibia vBMD (mg/cm^3), measured by pQCT (slice thickness 2.4mm, default voxel size of 0.5mm) at baseline, month 6, month 12, month 18, and month 24.
Additional variables by pQCT - tBMD Distal Femur | Baseline (0), Month 6, Month 12, Month 18, Month 24
  Percent change in distal femur trabecular BMD (tBMD) (mg/cm^3) will be measured by pQCT (slice thickness 2.4mm, default voxel size of 0.5mm) at baseline, month 6, month 12, month 18, and month 24.
Additional variables by pQCT - tBMD Proximal Tibia | Baseline (0), Month 6, Month 12, Month 18, Month 24
  Percent change in proximal tibia tBMD (mg/cm^3) will be measured by pQCT (slice thickness 2.4mm, default voxel size of 0.5mm) at baseline, month 6, month 12, month 18, and month 24.
Additional variables by pQCT - cortical BMD of the tibia (38% of the tibial length) | Baseline (0), Month 6, Month 12, Month 18, Month 24
  Percent change in cortical vBMD (mg/cm^3) will be measured by pQCT (slice thickness 2.4mm, default voxel size of 0.5mm) at baseline, month 6, month 12, month 18, and month 24.
Additional variables by pQCT - Distal Tibia Microarchitecture | Baseline (0), Month 6, Month 12, Month 18, Month 24
  Through the use of a custom software package (pQCT OsteoQ, Inglis Software Solutions Inc., Hamilton, ON) combined threshold-based and region-growing algorithms will be used to measure trabecular microarchitecture [trabecular separation (Tb.Sp), bone volume fraction (BV/TV), trabecular number (Tb.N), and trabecular thickness (Tb.Th)] at baseline, month 6, month 12, month 18, and month 24.
Additional variables by DXA - aBMD Distal Femur and Proximal Tibia (i.e. knee) | Baseline (0), Month 6, Month 12, Month 18, Month 24
  Percent change of regional BMD of the knee (e.g., distal femoral and proximal tibial epiphyses using the orthopedic knee software commercially available from GE Lunar). The starting point to acquire the knee is set on the tibia approximately 10 cm distal from the edge of the patella, with the scan field extending to the epiphysis and metaphysis of the distal femur. aBMD measurements will be taken at Baseline (0), Month 6, Month 12, Month 18, Month 24.
Additional variables by DXA - aBMD Hip | Baseline (0), Month 6, Month 12, Month 18, Month 24
  Percent change in aBMD of the hips (total dual dip and subregions) will be measured at Baseline (0), Month 6, Month 12, Month 18, Month 24. Accepted values for T-score and Z-scores of the hip will be utilized.
Biomarkers for Bone Resorption (CTx) | Baseline (0), Month 1, Month 3, Month 6, Month 12, Month 18, Month 24
  Change in levels of the circulating biochemical markers of bone resorption and formation before (baseline) and after initiating romosozumab therapy (1, 3, 6, and 12 months), and then after 6 and 12 months of denosumab administration will be measured. Levels of serum C-telopeptide (CTx) (ABclonal. 86 Cummings Park, Woburn, MA) will be measured as the biomarker of bone resorption.
Biomarkers for Bone Formation (osteocalcin, alkaline phosphatase, P1NP) | Baseline (0), Month 1, Month 3, Month 6, Month 12, Month 18, Month 24
  Change in levels of the circulating biochemical markers of bone resorption and formation before (baseline) and after initiating romosozumab therapy (1, 3, 6, and 12 months), and then after 6 and 12 months of denosumab administration will be measured. Serum osteocalcin (Alpco Diagnostics, Salem, NH), bone alkaline phosphatase (MyBiosource, Inc., San Diego, CA) and propeptide of type 1 procollagen (P1NP) (MyBiosource, Inc., San Diego, CA) will be measured as biomarkers of bone formation.
Calcium Metabolism Studies | Baseline (0), Month 1, Month 3, Month 6, Month 12, Month 18, Month 24
  Serum total and ionized calcium concentration, 24-hour urine calcium, 25 OH-vitamin D level (DiaSorin Inc. Stillwater, MN), 1,25 (OH)2-vitamin D level (Quest Diagnostics), and intact PTH level (ALPCO Diagnostics, Salem, NH) will be measured.The serum 25 OH-vitamin D level will be measured at baseline and 12 and 24 months; more frequent measurement will be performed, if indicated. Serum total and ionized calcium concentrations will be measured at baseline, 1, 3 months, and at 6-month intervals until month 24.
General Endocrine Studies | Baseline (0), Month 12, Month 24
  Serum thyroid function (T3, T4, & TSH; DiaSorin Inc. Stillwater, MN) will be determined by kit assay.
Additional variables by pQCT - Distal Tibia Microarchitecture | Baseline (0), Month 6, Month 12, Month 18, Month 24
  Through the use of a custom software package (pQCT OsteoQ, Inglis Software Solutions Inc., Hamilton, ON) combined threshold-based and region-growing algorithms will be used to bone volume fraction (BV/TV)at baseline, month 6, month 12, month 18, and month 24.
Additional variables by pQCT - Distal Tibia Microarchitecture | Baseline (0), Month 6, Month 12, Month 18, Month 24
  Through the use of a custom software package (pQCT OsteoQ, Inglis Software Solutions Inc., Hamilton, ON) combined threshold-based and region-growing algorithms will be used to measure trabecular number (Tb.N) at baseline, month 6, month 12, month 18, and month 24.
Additional variables by pQCT - Distal Tibia Microarchitecture | Baseline (0), Month 6, Month 12, Month 18, Month 24
  Through the use of a custom software package (pQCT OsteoQ, Inglis Software Solutions Inc., Hamilton, ON) combined threshold-based and region-growing algorithms will be used to measure trabecular thickness (Tb.Th)at baseline, month 6, month 12, month 18, and month 24.
Calcium Metabolism Studies | Baseline (0), Month 1, Month 3, Month 6, Month 12, Month 18, Month 24
  Serum ionized calcium concentration will be measured at baseline, months 1, 3, 6, 12, 18, and 24.
Calcium Metabolism Studies | Baseline (0), Month 1, Month 3, Month 6, Month 12, Month 18, Month 24
  24-hour urine calcium will be measured at baseline, months 1, 3, 6, 12, 18, and 24.
Calcium Metabolism Studies | Baseline (0), Month 1, Month 3, Month 6, Month 12, Month 18, Month 24
  25 OH-vitamin D levels (DiaSorin Inc. Stillwater, MN) will be measured at baseline and 12 and 24 months; more frequent measurement will be performed, if indicated.
Calcium Metabolism Studies | Baseline (0), Month 1, Month 3, Month 6, Month 12, Month 18, Month 24
  1,25 (OH)2-vitamin D level (Quest Diagnostics), will be measured at baseline and 12 and 24 months; more frequent measurement will be performed, if indicated.
Calcium Metabolism Studies | Baseline (0), Month 1, Month 3, Month 6, Month 12, Month 18, Month 24
  Intact PTH level (ALPCO Diagnostics, Salem, NH) will be measured at Baseline (0), Month 1, Month 3, Month 6, Month 12, Month 18, Month 24
General Endocrine Studies | Baseline (0), Month 12, Month 24
  Serum cortisol will be measured by kit assay (MP Biomedicals, Orangeburg, NY).
General Endocrine Studies | Baseline (0), Month 12, Month 24
  Serum total testosterone (T) will be determined by kit assay (MP Biomedicals, Orangeburg, NY).
General Endocrine Studies | Baseline (0), Month 12, Month 24
  Serum free testosterone (calculated from total T, albumin and SHBG) will be measured by kit assay (MP Biomedicals, Orangeburg, NY).
General Endocrine Studies | Baseline (0), Month 12, Month 24
  Serum estradiol (E2) will be measured by kit assay (MP Biomedicals, Orangeburg, NY).
General Endocrine Studies | Baseline (0), Month 12, Month 24
  Serum growth hormone (GH) will be measured by kit assay (MP Biomedicals, Orangeburg, NY).
General Endocrine Studies | Baseline (0), Month 12, Month 24
  Serum insulin-like growth factor-1 (IGF-I) will be measured by kit assay (ALPCO Diagnostics, Salem, NH).
Biomarkers for Bone Formation | Baseline (0), Month 1, Month 3, Month 6, Month 12, Month 18, Month 24
  Change in levels of bone alkaline phosphatase (MyBiosource, Inc., San Diego, CA) at baseline, month 1, month 3, month 6, month 12, month 18, and month 24.
Biomarkers for Bone Formation | Baseline (0), Month 1, Month 3, Month 6, Month 12, Month 18, Month 24
  Change in levels of propeptide of type 1 procollagen (P1NP) (MyBiosource, Inc., San Diego, CA) at baseline, month 1, month 3, month 6, month 12, month 18, and month 24.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Cardozo, MD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (2):
- United States (2):
  - Kessler Institute for Rehabilitation, West Orange, New Jersey
  - James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

DOCUMENTS (1):
  • Informed Consent Form (2023-12-27): https://cdn.clinicaltrials.gov/large-docs/57/NCT04232657/ICF_000.pdf